CLINICAL TRIAL: NCT07148271
Title: A Prospective Study Evaluating the Effects of a Dietary Supplement Product on Gut Microbiota and Ocular Surface Parameters in Patients With Dry Eye Disease
Brief Title: Effect of a Dietary Supplement on Gut Microbiota and Ocular Surface Outcomes in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varol TUNALI (Industry)
Collaborators: Istanbul Medipol University Hospital (Other); Liv Hospital (Ulus) (Unknown)
Responsible Party: Sponsor-Investigator, Varol TUNALI, Doctor, ENBIOSIS BIOTECHNOLOGIES
Organization: ENBIOSIS BIOTECHNOLOGIES (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-202.3.02-444
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye; Age-Related Macular Degeneration (AMD); Age-related Macular Degeneration (ARMD)
MeSH Terms: conditions — Dry Eye Syndromes; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement Product

INTERVENTIONS:
Dietary Supplement: Dietary Supplement Product — Participants will receive a dietary supplement product administered orally once daily for 8 weeks. The supplement is provided in capsule form and taken with water. The intervention is designed to modulate gut microbiota composition and diversity, with the potential to influence ocular surface outcomes in patients with dry eye disease. The regimen will be self-administered at home, with adherence monitored at study visits. Stool samples will be collected at baseline and week 8 for metagenomic sequencing, and ocular surface parameters will be assessed at the same time points. Safety will be evaluated by monitoring for adverse events throughout the intervention period.

SUMMARY:
This prospective clinical study investigates whether a dietary supplement product can modulate the gut microbiota and improve ocular surface outcomes in patients with dry eye disease. Participants will be recruited from Istanbul Medipol University Hospital (Department of Ophthalmology) and Liv Hospitals (Vadi Istanbul and Ulus). Each participant will receive the dietary supplement product for 8 weeks. Gut microbiota analyses will be conducted at baseline and week 8. Ocular surface assessments including Schirmer test and invasive tear breakup time (TBUT) will be performed at baseline and week 8.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifactorial ocular surface disorder characterized by chronic tear film instability, hyperosmolarity, and ocular surface inflammation. It represents one of the most common reasons for ophthalmology consultations worldwide and has a profound impact on patient quality of life. Conventional treatment approaches primarily target symptoms and tear film supplementation, but disease-modifying interventions remain limited.

Emerging evidence suggests that the gut microbiota exerts systemic immunomodulatory effects, influencing diseases beyond the gastrointestinal tract, including ocular conditions. Dysbiosis has been implicated in autoimmune, metabolic, and inflammatory disorders, and a growing body of literature indicates that the gut-eye axis may play a role in the pathogenesis of DED. Specific microbiota-derived metabolites, microbial antigens, and immune pathways are believed to modulate ocular surface inflammation and tear film stability. This provides a strong rationale for exploring microbiome-targeted interventions in DED.

This single-arm, prospective interventional trial investigates the impact of an 8-week course of a defined dietary supplement product on gut microbiota composition and diversity, alongside established ocular surface clinical endpoints. Participants will be recruited from Istanbul Medipol University Hospital (Department of Ophthalmology) and Liv Hospitals (Vadi Istanbul and Ulus). All enrolled patients will receive the dietary supplement once daily for the study duration.

Microbiome assessment: Stool samples will be collected at baseline and at week 8, with DNA extraction followed by metagenomic sequencing. Microbiota analysis will focus on alpha diversity (e.g., Shannon index) and taxonomic/functional profiling to detect shifts in microbial composition associated with the intervention.

Ophthalmological assessment: Clinical evaluations will be performed at baseline and at week 8, including the Schirmer test, invasive tear breakup time (TBUT), Ocular Surface Disease Index (OSDI), and Dry Eye Scoring System (DESS). These standardized measures provide quantitative and qualitative assessment of tear production, stability, and patient-reported symptoms.

Safety and adherence: Safety monitoring will include the recording of adverse events throughout the trial, with particular attention to potential gastrointestinal or ocular side effects. Adherence will be assessed through participant reporting and calculation of percentage of doses taken.

Statistical considerations: Data will be analyzed using SPSS v22.0. Non-parametric tests (Mann-Whitney U for between-group and Wilcoxon signed-rank for within-group comparisons, where applicable) will be employed, as clinical data are expected to be non-normally distributed. Descriptive statistics will summarize adherence and adverse events.

This study aims to provide mechanistic insights into the gut-eye axis by linking microbiome modulation with ocular surface outcomes. Although exploratory in design, the findings may lay the groundwork for future randomized controlled trials evaluating microbiome-targeted interventions as adjunctive therapy for DED.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dry eye disease.
* Age 18-65 years.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Current restrictive diet (ketogenic, elimination, prolonged fasting, etc.).
* Colonoscopy or systemic antibiotic use within the past 4 weeks.
* Use of probiotic, prebiotic, or fecal microbiota-related products within the past 4 weeks.
* Other systemic or ocular conditions that could interfere with study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test Score | From enrollment to the end of treatment at 8 weeks
  Tear production will be assessed using the Schirmer Test without anesthesia at baseline and at week 8. Standardized Schirmer paper strips will be placed in the lower eyelid, and the length of strip wetting (measured in millimeters) will be recorded after 5 minutes.
  The Schirmer Test yields values ranging from 0 mm (no tear production) to approximately 35 mm (normal/high tear production) over 5 minutes. Higher values represent better tear production, while values <10 mm/5 min are commonly associated with clinically significant dry eye disease.
  The primary endpoint is the mean change in Schirmer Test score from baseline to week 8.

SECONDARY OUTCOMES:
Change in Tear Breakup Time (TBUT, invasive) | From enrollment to the end of treatment at 8 weeks
  Tear film stability will be assessed at baseline and week 8 using the Fluorescein Tear Breakup Time Test. After instillation of fluorescein dye into the tear film, the time (in seconds) between a complete blink and the appearance of the first dry spot on the cornea will be recorded. TBUT values typically range from 0 seconds (immediate breakup, very unstable tear film) to >10 seconds (normal tear film stability). Shorter TBUT values indicate worse tear film stability and more severe dry eye disease.
Change in Ocular Surface Disease Index (OSDI) | From enrollment to the end of treatment at 8 weeks
  The Ocular Surface Disease Index (OSDI) questionnaire will be administered at baseline and week 8. The OSDI consists of 12 items evaluating ocular discomfort, vision-related function, and environmental triggers. Scores range from 0 to 100, where 0 indicates no symptoms and 100 indicates the most severe dry eye symptoms. Higher scores represent worse outcomes.
Change in Dry Eye Scoring System (DESS) | From enrollment to the end of treatment at 8 weeks
  The Dry Eye Scoring System (DESS) will be administered at baseline and week 8 to evaluate the severity and frequency of dry eye symptoms. Scores range from 0 (no symptoms) to 44 (maximum severity and frequency of symptoms). Higher scores represent worse outcomes.
Change in gut microbiota diversity (Shannon index) | From enrollment to the end of treatment at 8 weeks
  Stool samples will be collected at baseline and week 8 for metagenomic sequencing. Alpha diversity will be measured using the Shannon Diversity Index, which accounts for both richness and evenness of microbial communities. Shannon index values are non-negative and typically range from 0 (no diversity) to approximately 5-6 (very high diversity in complex communities). Higher Shannon index values represent greater microbial diversity, which is generally considered a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Varol TUNALI, Dr., Principal Investigator — Celal Bayar University Faculty of Medicine Parasitology Department
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study (after de-identification) will be made available to researchers upon reasonable request. Data to be shared include demographic variables, outcome measures (ocular surface parameters, microbiome sequencing data, and safety/adherence data), and relevant baseline characteristics. A data dictionary will be provided to allow full interpretation.
  The data will become available following publication of the primary study results and will be accessible for a period of 5 years thereafter. Researchers may request access by contacting the principal investigator. Requests will be evaluated on a case-by-case basis, and data will be shared for scientifically valid proposals in accordance with ethical approvals and data protection regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: May 2026-May 2031